CLINICAL TRIAL: NCT05543070
Title: Low-dose Radiotherapy in Indolent Lymphoma：A Multi-center Phase II Study
Brief Title: Low-dose Radiotherapy in iNHL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Shanxi Province Cancer Hospital (Other); Beijing Tongren Hospital (Other); Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Shunan Qi, Associated Prof. in the radiation oncology department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCG-iNHL-01
Record Dates: First submitted 2022-09-08; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Indolent Lymphoma; Low-dose Radiotherapy
Keywords: indolent lymphoma; low-dose radiotherapy
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-dose Radiotherapy (Experimental): Involved-site radiotherapy (3 Gy*4f) in one week
  Interventions: Radiation: Low-dose radiotherapy

INTERVENTIONS:
Radiation: Low-dose radiotherapy — Electron Beam/3D-CRT/IMRT/VMAT

SUMMARY:
The current study is a phase II multi-center single arm trial to evaluate the efficacy and safety of low-dose radiotherapy (3 Gy*4f) in indolent lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathology proved iNHL
* ECOG PS ≤3
* Signed Informed consent

Exclusion Criteria:

* History of radiotherapy at the same site
* Primary malignant lymphoma of the gastrointestinal tract
* CTV (Clinical Target Volume)>500ml
* Others that researchers consider inappropriate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical complete response after radiotherapy | 6-month after radiotherapy
  complete resolution of disease in imaging or biopsy after low-dose radiotherapy

SECONDARY OUTCOMES:
Overall response rate after radiotherapy | 6-month after radiotherapy
  complete or partial resolution of disease in imaging or biopsy after low-dose radiotherapy
Progression-free survival rate at year 2 after enrollment, 2y-PFS | 2-year
  From enrollment to any disease progression or death
Local control rate at year 2 after enrollment, 2y-LCR | 2-year
  From enrollment to any local disease progression or death
Rate of acute toxicity (any and above grade 3) | From enrollment to 3 months after treatment
  toxicities according to CTCAE criteria
Rate of late toxicity (any and above grade 3) | After 3 months of enrollment
  toxicities according to CTCAE criteria
Quality of Life change, QoL | 1/3/6/12/24 months after radiotherapy
  measurement basing on EORTC-QLQ-C30 tables

OTHER OUTCOMES:
Biomarkers to predict radiotherapy efficacy | baseline/through study completion, an average of 1 year
  potential biomarkers in baseline tumor samples and blood samples
Conjunctival microbiota | baseline/4 fractions/1/3/6/12/24 months after radiotherapy
  DNA samples from ocular adnexal extranodal MALT lymphoma patients' conjunctiva

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From: 6 months after publication. To: 5 years after publication
Access Criteria: Will share data with the PIs who had specific study plan in tumor sequencing analysis

REFERENCES:
- [Derived] Wang XY, Zhang XM, Wang L, Gao LR, Chen K, Feng XL, Rao W, Zheng R, Wu YP, Song YW, Fang H, Chen B, Jin J, Liu YP, Jing H, Tang Y, Zhang WW, Zhai YR, Lu NN, Li N, Xia CF, Wang SL, Liu X, Li YX, Qi SN. Low-dose moderate hypofractionated radiotherapy for indolent non-Hodgkin lymphoma: a multicentre, single-arm, phase 2 trial. Lancet Haematol. 2025 Jun;12(6):e442-e450. doi: 10.1016/S2352-3026(25)00071-7. Epub 2025 May 2. PMID 40324445
- [Derived] Gao LR, Wang X, Xia C, Song YW, Wang L, Li X, Yang Y, Cao JZ, Chen K, Zhong QZ, Gao Y, Zhou SY, Feng XL, Wang X, Li YX, Qi SN. Multicenter phase II study of moderate low-dose radiotherapy in indolent non-Hodgkin lymphoma: CLCG-iNHL-01 protocol. Future Oncol. 2024 Jan;20(2):71-81. doi: 10.2217/fon-2023-0761. Epub 2024 Jan 5. PMID 38179936